CLINICAL TRIAL: NCT03889470
Title: A Randomized Comparison of Nitroglycerin Versus Placebo as Spasmolytic Regimen to Prevent Moderate to Severe Radial Artery Spasm in Radial Center
Brief Title: Nitroglycerin as Spasmolytic Regimen for RAS Prevention in Radial Center
Acronym: NORAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hermina Heart Center Kemayoran (Other)
Responsible Party: Principal Investigator, Surya Dharma, MD, PhD, MD, PhD, Hermina Heart Center Kemayoran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HerminaHCKRAS
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Radial Artery Injury
Keywords: transradial catheterisation; radial artery spasm
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: NTG vs Placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 200 microgram NTG (Active Comparator): 200 microgram NTG through the radial sheath
  Interventions: Drug: NTG 1 MG/ML Injectable Solution
- Saline (Placebo Comparator): Saline infusion through the radial sheath
  Interventions: Drug: NTG 1 MG/ML Injectable Solution

INTERVENTIONS:
Drug: NTG 1 MG/ML Injectable Solution — administered after sheath placement
  Other Names: Nitroglycerin

SUMMARY:
The investigators will investigate whether administration of Nitroglycerin (NTG) as spasmolytic regimen reduces the incidence of moderate to severe radial artery spasm (RAS) in patients undergoing transradial catheterization in radial center.

DETAILED DESCRIPTION:
Patients will be randomized to receive either 200 microgram NTG or placebo (saline) at the beginning of the procedure soon after radial sheath placement. The operators will be blinded to both assignment. The primary outcome is the incidence of moderate to severe RAS evaluated by the operators during the radial procedure.

Both NTG and placebo will be administered using an identical syringe to keep the operators blinded to the treatment allocation. Radial angiogram is mandatory to measure the diameter of both radial and ulnar arteries. Doppler ultrasound of the radial artery will be examined at the day after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing transradial catheterisation using proximal radial artery puncture technique

Exclusion Criteria:

* Blood pressure <100 mmHg
* Refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-31 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of Moderate to severe radial artery spasm | During the index procedure
  arm pain associated with catheter manipulation (RAS grade 2 to 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Hermina Heart Center, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No